CLINICAL TRIAL: NCT02138032
Title: Effects of Message Content on Intention to Quit Smoking in Smokers With Peripheral Artery Disease - a Randomised Controlled Trial
Brief Title: Effects of Message Content on Intention to Quit Smoking
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Student study which ended at the end of their course.
Sponsor: University of Stirling (Other)
Collaborators: NHS Forth Valley (Other Government)
Responsible Party: Principal Investigator, Maggie Cunningham, Lecturer Health Psychology, University of Stirling
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CUNN-001-RCT
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Peripheral Artery Disease
Keywords: message framing; smoking cessation; peripheral artery disease
MeSH Terms: conditions — Peripheral Arterial Disease; Smoking Cessation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gains Framed Message (Experimental): gains framed visual fridge magnet and information sheet about smoking cessation (benefits of quitting smoking)
  Interventions: Behavioral: Gains Framed Message
- Loss Framed Message (Experimental): loss framed visual fridge magnet and information sheet about smoking cessation (losses of continued smoking)
  Interventions: Behavioral: Loss Framed Message

INTERVENTIONS:
Behavioral: Gains Framed Message
  Arms: Gains Framed Message
Behavioral: Loss Framed Message
  Arms: Loss Framed Message

SUMMARY:
Message framing involves "the presentation of choice alternatives, either in a positive or negative manner" (Huber, Neale, & Northcraft, 1987; p.137). Positively framed health messages contain potential gains of participating/refraining in specific health behaviour. Alternatively, negatively framed health messages contain potential losses of participating/refraining in specific health behaviour (Verlhiac, Chappe, & Meyer, 2011). The primary aim and rationale of this study will be to investigate which type of framing has the greatest effect on intentions to quit smoking in patients with vascular arterial disease. The secondary aim is to investigate what other factors may have an effect on intention to quit and also what factors play a part in a patient's intention to quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral Artery Disease
* daily smoker

Exclusion Criteria:

* psychiatric illness or those who are not literate in English will be excluded from the study as informed consent cannot be obtained. Also, patients who are already participating in any other research involving smoking cessation will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Intention to quit smoking | up to 3 weeks
  Intention to quit smoking will be assessed by measuring the strength of the individual's intention with a mean score being calculated from the 3 questions asked. This will generate a score between 1 and 7 with a higher score indicating a higher intention to quit smoking. This measure has been used and reviewed in previous research (Francis et al, 2004).

SECONDARY OUTCOMES:
Stage of Change - smoking cessation | baseline and 3 weeks
  Secondly, the Stage of Change (SOC) of intention will be measured, with higher scores indicating a greater intention to quit smoking. The corresponding scores will identify the SOC (1 =pre-contemplation, 2 = contemplation, 3 = preparation, 4 = action). This measure has been adapted from a previous study which investigated stages of change in relation to smoking cessation (Fathelrahman et al. 2009).
Nicotine Dependence | Baseline and 3 weeks
  Nicotine dependency will be measured using the standardised Fagerstrom Test for Nicotine Dependence (FTNP: Heatherton, Kozlowski, Frecker, & Fagerstrom, 1991)
Outcome expectancy beliefs | Baseline and 3 weeks
  Expectancy beliefs will be measured using a 10-item questionnaire which has been adapted from the Health Action Process Approach (HAPA) assessment tools (Schwarzer, 2007) by making the questions relevant to the specific patient group. The questionnaire is comprised of two sub-scales: positive outcome expectancies (items 1, 3, 4, 6, 9) and negative outcome expectancies (items 2, 5, 7, 8, 10). Each subscale sum scores will range from 5-20.
Self efficacy | Baseline and 3 weeks
  Self-efficacy to quit smoking will be measured using a 10-item scale which has been previously used in a study investigating self-efficacy influences on the effects of framing in smoking cessation (Riet, Ruiter, Werrij, & de Vries, 2008). Sum scores will range from 10 to 70 with higher scores indicating greater self-efficacy to quit smoking.
Risk Perception | baseline and 3 weeks
  Risk perception of smoking will be measured using a 5-item questionnaire. The items are similar to that used in a previous study (Clarke and Aish, 2002), however the questions have been adapted to increase the relevance for vascular arterial patients. Sum scores will range from 5-35 with higher scores indicating a greater risk perception in regards to smoking.
Health locus of control | baseline and 3 weeks
  Health locus of control will be measured using the Multidimensional Health Locus of Control Scale - Form C (MHLC; Wallston, Stein & Smith, 1994).

CONTACTS AND LOCATIONS:
Locations (1):
- Forth Valley Royal Hospital, Larbert, Falkirk, United Kingdom